CLINICAL TRIAL: NCT05272969
Title: Pompe & Pain - Observational Study to Assess Musculoskeletal Pain in Late-onset Pompe Disease (LOPD)
Brief Title: Pompe & Pain - Study to Assess Nociceptive Pain in Adult Patients With Pompe Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Prof. Dr. Benedikt Schoser, Professor of Neurology, LMU Klinikum
Other Study IDs: Pompe&Pain
Record Dates: First submitted 2022-01-28; First posted 2022-03-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Pompe Disease (Late-onset); Inclusion Body Myositis; Spinal Muscular Atrophy Type 3; FSHD
MeSH Terms: conditions — Glycogen Storage Disease Type II; Myositis, Inclusion Body; Spinal Muscular Atrophies of Childhood | interventions — Walk Test; Vital Signs; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Polymorphisms of ACE and ACTN3. Upon additional informed consent, exome sequencing will be performed in a second step to assess whether polymorphisms or pathogenic mutations in genes that are associated with chronic pain syndromes contribute to increased pain. The selection of the genes is based on the Human Phenotype Ontology (HPO) search terms "myalgia", "muscle pain", "chronic pain", "musculoskeletal pain", "pain", and "nociceptive pain".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LOPD group: 50 Patients with genetically confirmed late-onset Pompe disease.
  Interventions: Diagnostic Test: Beck depression inventory fast screen (Questionnaire); Diagnostic Test: Brief Pain Inventory (BPI) (Questionnaire); Diagnostic Test: German Pain Inventory (Questionnaire); Diagnostic Test: Fatigue Severity and Disability Scale (FSS) (Questionnaire); Diagnostic Test: Rotterdam Handicap Scale (RHS) (Questionnaire); Diagnostic Test: R-PAct (Questionnaire); Diagnostic Test: Quick Motor Function Test; Diagnostic Test: Handheld Dynamometry (HHD); Diagnostic Test: Six-minute walk test (6MWT); Diagnostic Test: Pressure pain threshold; Diagnostic Test: Muscle ultrasound; Diagnostic Test: Vital signs; Diagnostic Test: Borg Scale; Diagnostic Test: Laboratory assessment: Creatine kinase; Diagnostic Test: Laboratory assessment: Vitamin D Level; Diagnostic Test: Laboratory assessment: calcium; Diagnostic Test: Laboratory assessment: magnesium; Diagnostic Test: Laboratory assessment: phosphate; Genetic: Genetic test: ACE polymorphism; Genetic: Genetic test: ACTN3 polymorphism; Genetic: Blood draw for optional genetic exome sequencing
- Control group: 15 Patients with histologically confirmed inclusion body myositis (IBM), 15 patients with genetically confirmed spinal muscular atrophy type 3 (SMA3) and 15 patients with genetically confirmed facio-scapulo-humeral muscle dystrophy (FSHD) will serve as a control group.
  Interventions: Diagnostic Test: Beck depression inventory fast screen (Questionnaire); Diagnostic Test: Brief Pain Inventory (BPI) (Questionnaire); Diagnostic Test: German Pain Inventory (Questionnaire); Diagnostic Test: Fatigue Severity and Disability Scale (FSS) (Questionnaire); Diagnostic Test: Rotterdam Handicap Scale (RHS) (Questionnaire); Diagnostic Test: R-PAct (Questionnaire); Diagnostic Test: Quick Motor Function Test; Diagnostic Test: Handheld Dynamometry (HHD); Diagnostic Test: Six-minute walk test (6MWT); Diagnostic Test: Pressure pain threshold; Diagnostic Test: Muscle ultrasound; Diagnostic Test: Vital signs; Diagnostic Test: Borg Scale; Diagnostic Test: Laboratory assessment: Creatine kinase; Diagnostic Test: Laboratory assessment: Vitamin D Level; Diagnostic Test: Laboratory assessment: calcium; Diagnostic Test: Laboratory assessment: magnesium; Diagnostic Test: Laboratory assessment: phosphate; Genetic: Genetic test: ACE polymorphism; Genetic: Genetic test: ACTN3 polymorphism; Genetic: Blood draw for optional genetic exome sequencing

INTERVENTIONS:
Diagnostic Test: Beck depression inventory fast screen (Questionnaire) — Beck depression inventory fast screen questionnaire to detect severe depression for eligibility.
Diagnostic Test: Brief Pain Inventory (BPI) (Questionnaire) — Validated questionnaire for pain.
Diagnostic Test: German Pain Inventory (Questionnaire) — German Pain Inventory questionnaire for evaluation of pain. Module A, abbreviated questions of module S (sociodemographic questions S1, S2, S3, S4, S5 and S8) and module L (quality of life) and V (therapies) will be used.
  Other Names: Deutscher Schmerzfragebogen (DSF)
Diagnostic Test: Fatigue Severity and Disability Scale (FSS) (Questionnaire) — Validated questionnaire for perceived fatigue
Diagnostic Test: Rotterdam Handicap Scale (RHS) (Questionnaire) — validated questionnaire to assess a patient's functional ability and level of handicap
Diagnostic Test: R-PAct (Questionnaire) — The R-PAct scale is designed specifically for Pompe disease, which consists of 18 items addressing daily life activities with three response options.
Diagnostic Test: Quick Motor Function Test — An evaluator observes the performance of a patient and scores the items separately on a 5-point ordinal scale (ranging from 0 to 4). A total score is obtained by adding the scores of all items and ranges between 0 and 64 points.
Diagnostic Test: Handheld Dynamometry (HHD) — To ensure a high level of objective measurement, muscle strength will also be assessed by handheld dynamometry. The following muscle groups will be tested: Arm abduction, elbow flexion, elbow extension, hip flexion, hip extension, knee extension, knee flexion, foot extension, foot flexion.
Diagnostic Test: Six-minute walk test (6MWT) — It is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. If a six-minute-walk-test was performed within the last 3 months within the routine treatment, no additional test will be performed and the distance walked in meters as well as borg scale will be recorded in the study CRF, including the date of the assessment. If not performed within the last six months, a six-minute-walk test will be performed once.
Diagnostic Test: Pressure pain threshold — For diagnosis of myofascial pain, pressure algometers are designed and conventionally used to measure deep pressure pain thresholds or tenderness resistance (Park, Kim et al. 2011), and the reliability of pressure pain thresholds according to raters or measurement frequencies has been proven to be relatively high (Chung, Um et al. 1992). The threshold is then determined as the arithmetic mean of the 3 series (in kPa). The measurement will be stopped immediately as the patient feels sensations of "burning", "stinging", "drilling" or "aching. Pressure algometry measurements will be performed on the trapezius, deltoid and supraspinatus muscles, the rectus femoris muscles, and the tibialis anterior muscles.
Diagnostic Test: Muscle ultrasound — Muscle ultrasound is an ideal imaging modality that allows for atraumatic, noninvasive, radiation-free point-of-care neuromuscular imaging. Muscular diseases are typically associated with an increase in the echogenicity from the muscle substance, distal attenuation of muscle echo and a corresponding loss of bone echo. A measurement on both sides deltoid, biceps and triceps brachii muscle, quadriceps femoris muscle, tibialis anterior muscle, rectus abdominis muscle and paravertebral muscles of cervical (C5-7), thoracic (Th4-6) and lumbar (L4-5) muscles. Muscle tissue alterations will be classified using the Heckmatt scale I-IV, describing muscle echogenicity. For muscle ultrasound, a linear 17MHz probe will be used. The muscle ultrasound assessment usually takes 15-20 minutes.
Diagnostic Test: Vital signs — Vital signs (blood pressure, heart rate, respiratory rate) will be measured before and after the six-Minute-Walk-Test (6MWT).
Diagnostic Test: Borg Scale — The Borg scale will be assessed, which is a self-reported questionnaire designed to subjectively assess dyspnea and exertion during activity (Borg 1982). The Borg scale rates dyspnea on a scale of 0 to 10 incorporating nonlinear spacing of verbal descriptors of the level of intensity of dyspnea. A higher Borg score indicates more severe dyspnea. The Borg scale will be administered before starting the 6MWT (≤ 5 minutes) and after completing the 6MWT (≤ 5 minutes).
Diagnostic Test: Laboratory assessment: Creatine kinase — CK-Level assessment in peripheral blood (peripheral venous blood draw)
Diagnostic Test: Laboratory assessment: Vitamin D Level — Vitamin D Level in peripheral blood (peripheral venous blood draw)
Diagnostic Test: Laboratory assessment: calcium — calcium level in peripheral blood (peripheral venous blood draw)
Diagnostic Test: Laboratory assessment: magnesium — magnesium level in peripheral blood (peripheral venous blood draw)
Diagnostic Test: Laboratory assessment: phosphate — phosphate level in peripheral blood (peripheral venous blood draw)
Genetic: Genetic test: ACE polymorphism — peripheral venous blood draw for genetic analysis of ACE polymorphism
Genetic: Genetic test: ACTN3 polymorphism — peripheral venous blood draw for genetic analysis of ACTN3 polymorphism
Genetic: Blood draw for optional genetic exome sequencing — Optionally, upon additional informed consent, exome sequencing from peripheral blood will be performed in a second step to assess whether polymorphisms or pathogenic mutations in genes that are associated with chronic pain syndromes contribute to increased pain. This analysis will be performed collectively after enrollment is complete by the Genetikum Neu-Ulm. The selection of the genes is based on the Human Phenotype Ontology (HPO) search terms "myalgia", "muscle pain", "chronic pain", "musculoskeletal pain", "pain", and "nociceptive pain".

SUMMARY:
The primary aim of this nationwide, explorative, cross-sectional study in Germany is to characterize the prevalence, severity and quality of musculoskeletal pain in adult patients with late-onset Pompe disease (LOPD). The secondary objectives are to evaluate whether muscle pain is associated with muscle function, to assess whether muscle pain is associated with alterations of muscle tissue, and whether vitamin D metabolism and polymorphisms of ACE and ACTN3 genes may contribute to an increased level of perceived musculoskeletal pain. In a second step, exome sequencing of genes associated with musculoskeletal pain will be analyzed. Results of LOPD patients will be compared to patients with neuromuscular disorders with a similar distribution of muscle weakness and/or musculoskeletal pain.

DETAILED DESCRIPTION:
In this nationwide, explorative, cross-sectional study in Germany, approx. 50 patients with genetically confirmed late-onset Pompe disease (LOPD) will be included into the study. In addition, 15 Patients with histologically confirmed inclusion body myositis (IBM), 15 patients with genetically confirmed spinal muscular atrophy type 3 (SMA3) and 15 patients with genetically confirmed facio-scapulo-humeral muscle dystrophy (FSHD) will serve as a control group. The duration of patient recruitment will be around 18 months. The primary aim is to characterize the prevalence, severity and quality of musculoskeletal pain in adult patients with late-onset Pompe disease (LOPD). The secondary objectives are to evaluate whether muscle pain is associated with muscle function, measured by quantitative muscle testing and pressure pain threshold (PPT), to assess whether muscle pain is associated with alterations of muscle tissue, measured by muscle ultrasound and whether vitamin D metabolism and polymorphisms of ACE and ACTN3 genes may contribute to an increased level of perceived musculoskeletal pain. In a second step, exome sequencing of genes associated with musculoskeletal pain will be analyzed. Results of LOPD patients will be compared to patients with neuromuscular disorders with a similar distribution of muscle weakness and/or musculoskeletal pain.

After screening of 120 patients, approximately 50 patients with late-onset Pompe disease, 15 patients with IBM, 15 patients with FSHD and 15 patients with SMA3, who meet all eligibility criteria, will be enrolled in the study. All patients will be required to attend once at a study site to perform all study-related procedures. The study procedures will take approx. 3 hours.

Demographic and disease-related data (age, gender, weight, height, diagnosis, a historical genetic test results and/or muscle biopsy results, age at onset of symptoms, age at diagnosis, severity and distribution of muscle weakness, prior and concomitant medication, medical history, ventilation status) will be obtained. Patients will fill out validated disease-related and quality-of-life questionnaires: Brief Pain Inventory, Rotterdam Handicap Scale, Fatigue Severity Scale, R-PAct, and German Pain Questionnaire. Patients will be asked to sketch regions of perceived musculoskeletal pain on a body figure, which is provided on a tablet or a paper version. The paper version will be scanned and regions of muscular pain will be digitally evaluated to develop a map of musculoskeletal pain regions. For this, a novel software will be used, provided by the Institute for Information Engineering, Wolfenbüttel.

Muscle strength will be assessed clinically by MRC grading (0-5), by quick motor function test (QMFT) and by dynamometry of selected muscles.

Pressure Pain Threshold (PPT) is defined as the minimum force applied which induces pain. Pressure algometry measurements will be performed to assess PPTs on the trapezius, deltoid and supraspinatus muscles, the rectus femoris muscles, and the tibialis anterior muscles. For muscle function and endurance, a six-minute walk test will be performed. If this test was performed within the last 3 months (e.g. for routine treatment/assessments), no new test will be performed and the last assessment will be documented (distance walked in meters, borg scale, vital parameters and date of assessment). In muscle ultrasound, alterations of muscle tissue will be evaluated in selected muscles of proximal muscles of upper and lower limbs, cervical, thoracic and lumbar vertebral muscles and rectus abdominis muscle. In laboratory assessments, polymorphisms of ACE and ACTN3 will be analyzed by molecular analysis. Levels of creatine kinase (CK) and Vitamin D, calcium, phosphate and magnesium will be analyzed. In a second step upon additional informed consent, blood samples will be analyzed by exome sequencing for mutations and variants in common genes associated with chronic pain syndromes.

ELIGIBILITY:
Inclusion Criteria: A patient must meet the following criteria to be eligible for this study:

1. The patient is willing and able to provide signed informed consent.
2. The patient is able and willing to perform study-related assessments.
3. A) The patient is ≥18 years of age with acid α-glucosidase [GAA] enzyme deficiency, confirmed by GAA gene mutation analysis, or B) The patient has a histologically confirmed diagnosis of inclusion body myositis (IBM), or a genetically confirmed spinal muscular atrophy type 3 (SMA3) or a genetically confirmed facio-scapulo-humeral muscle dystrophy (FSHD).

Exclusion Criteria: A patient who meets any of the following criteria will be excluded from this study.

1. The patient is participating in another clinical study or using an investigational treatment.
2. The patient, in the opinion of the Investigator, is unable to adhere to the requirements of the study.
3. The patient has currently a severe depression, assessed by the Beck depression inventory fast screen (BDI-FS) with a score ≥ 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After screening of 120 patients, approximately 50 patients with late-onset Pompe disease, 15 patients with IBM, 15 patients with FSHD and 15 patients with SMA3, who meet all eligibility criteria, will be enrolled in the study. All patients must be ≥ 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-09-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of musculoskeletal pain in LOPD patients | Only at baseline visit
  The primary aim of this nationwide, explorative, cross-sectional study in Germany is to characterize the prevalence of musculoskeletal pain in adult patients with late-onset Pompe disease (LOPD).

SECONDARY OUTCOMES:
Association between musculoskeletal pain and muscle function, assessed by Medical research council (MRC) grading (0-5) | Only at baseline visit
  Assessed by Medical research council (MRC) grading (0-5) of selected muscles: on both sides deltoid muscles, biceps brachii muscles, triceps brachii muscles, hip flexors, hip extensors, quadriceps femoris muscles, foot extensor and foot flexor muscles as well as axial muscles and neck flexors and extensors. A maximum score of 95 means no weakness, a minimum score of 0 means tetraplegia.
Association between musculoskeletal pain and muscle function, assessed by quick motor function test (QMFT) | Only at baseline visit
  Assessed by quick motor function test (QMFT). The QMFT is a clinical test. An evaluator assesses the performance of a patient and scores the items separately on a 5-point ordinal scale, ranging from 0 (not able) to 4 (normal performance). A total score is obtained by adding the scores of all items. The total score ranges between 0 and 64 points, a higher score means better performance.
Association between musculoskeletal pain and muscle function, assessed by Pressure Pain Threshold (PPT) | Only at baseline visit
  Assessed by Pressure Pain Threshold (PPT). Pressure algometry is defined as the minimum force applied which induces pain. Measurements will be performed on the trapezius, deltoid and supraspinatus muscles, the rectus femoris muscles, and the tibialis anterior muscles. The assessor places the pressure algometer on a site to be inspected in 3 series of slowly increasing stimulus (contact area 1cm2) intensities (0.5 kg/s, corresponding to ca. 50 kPa/s). A higher score means a higher pressure pain threshold. There is no cutoff or total score.
Association between musculoskeletal pain and alterations of muscles, assessed by muscle ultrasound | Only at baseline visit
  To assess whether musculoskeletal pain regions are associated with muscle tissue alteration, evaluated by muscle ultrasound, using the Heckmatt scale 1 (no alteration) to IV (dystrophic muscle). Lower scale means healthier muscle.
Association between musculoskeletal pain and Insertion-(I)-/Deletion-(D)-Polymorphisms of the ACE (angiotensin-converting enzyme; (ACE-I/D)) gene | Only at baseline visit
  ACE genotyping (angiotensin-converting enzyme I/D polymorphisms) to assess whether Insertion-(I)-/Deletion-(D)-Polymorphisms of the ACE gene are associated with musculoskeletal pain.
Association between musculoskeletal pain and R-/X-polymorphisms of the Alpha-Actinin-3 (ACTN3) gene | Only at baseline visit
  ACTN3 genotyping (Alpha-Actinin-3 R-/X-polymorphisms) to assess whether R-/X-Polymorphisms of the ACTN3 gene are associated with musculoskeletal pain.
Association between musculoskeletal pain and variants in defined genes, using exome sequencing | Only at baseline visit
  to assess whether polymorphisms or pathogenic mutations in genes that are associated with chronic pain syndromes contribute to nociceptive pain, using exome sequencing of selected genes.
Characterization of musculoskeletal pain (quality and severity) assessed by the German Pain Questionnaire | Only at baseline visit
  Characterization of quality and severity of musculoskeletal pain. The German Pain Questionnaire is a multidimensional questionnaire, based on several modules to characterize the quality of pain and consists of: demographic data, pain variables (e. g. pain sites, temporal characteristics, duration), pain associated symptoms, affective and sensory qualities of pain, pain-relieving and intensifying factors, previous pain treatment procedures, pain-related disability, comorbid conditions, social factors, and health-related quality of life. Module A, abbreviated questions of module S (sociodemographic questions S1, S2, S3, S4, S5 and S8) and module L (quality of life) and V (therapies) will be used. However, there is no total score that indicates e.g. lower or higher pain.
Characterization of musculoskeletal pain (quality and severity) assessed by the Brief Pain Inventory (BPI) | Only at baseline visit
  To assess the severity of pain and the impact of pain on daily functions. The two categories Pain Intensity and Pain Interference are rated by patients on a scale from 0-10, 10 being excruciating pain intensity and a complete interference in their life. There is no scoring algorithm, but "worst pain" or the arithmetic mean of the four severity items can be used as measures of pain severity; the arithmetic mean of the seven interference items can be used as a measure of pain interference.

OTHER OUTCOMES:
Assessment of Questionnaire: Beck depression inventory fast screen | Only at baseline visit
  Association between Depression and musculoskeletal pain. Participants are asked to select the statement that describes best their feeling during the past 2 weeks by choosing the answer of four graded statements describing symptoms of depression on a scale ranging from zero to 3. The BDI-FS is then scored by summing the ratings of each item. Zero means no depressive symptoms, whereas a cut-off score of four and above indicates a major depression.
Assessment of Questionnaire: Rotterdam Handicap Scale (RHS) | Only at baseline visit
  Questionnaire evaluation: characteristics of musculoskeletal pain associated with score in Rotterdam Handicap Scale (RHS). The RHS provides information about mobility but also physical independence, occupation, and social integration for patients with neuromuscular disorders. The RHS consists of nine questions on the topics mobility indoors, mobility outdoors, kitchen tasks, domestic tasks indoors, domestic tasks outdoors, leisure activities indoors, leisure activities outdoors, travelling, and work or study. The scores per item range from 1 ('unable to fulfil the task or activity') to 4 ('complete fulfilment of the task or activity'). The total score ranges from 9 ('unable to fulfil any task/activity') to 36 ('able to fulfil all applicable tasks or activities').
Assessment of Questionnaire: R-Pact | Only at baseline visit
  The Rasch-built Pompe-specific activity (R-PAct) is a subject-reported disease-specific 18-item questionnaire using Rasch analysis specifically suited to quantify activity limitations, ranging from unable to perform daily life activities (0) to able to perform without difficulty (2) in patients with Pompe disease. A lower score indicates a higher limitation in activity of daily life.
Assessment of Questionnaire: Fatigue Severity and Disability Scale (FSS) | Only at baseline visit
  Questionnaire evaluation: characteristics of musculoskeletal pain associated with score in Fatigue Severity and Disability Scale (FSS). The Fatigue Severity Scale is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. The items are scored on a 7 point scale with 1=strongly disagree and 7=strongly agree. The minimum score=9 and maximum score possible=63. Higher the score=greater fatigue severity.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Wenninger, PD Dr. med., Principal Investigator — Study Principal Investigator
Locations (1):
- Friedrich-Baur-Institute, Dep. of Neurology Klinikum der Universitaet Muenchen, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No